CLINICAL TRIAL: NCT00324181
Title: Psychopathology of Normal-tension Glaucoma in Hong Kong Chinese Out-patient
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Dexter Yu-lung LEUNG/ Honorary Clinical Assistant Professor, DOVS, CUHK
Other Study IDs: CRE-2006.060
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Glaucoma
Keywords: normal-tension glaucoma; psychopathology; Hong Kong
MeSH Terms: conditions — Glaucoma; Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It is suggested the pathogenesis of normal-tension glaucoma (NTG) involves vascular dysregulation. In the past studies, it is well documented that many physical problems related to vascular dysregulation, such as angina pectoris (Friedman M et al 1974; Russek HI et al 1976), migraine (Diener HC et al 1994), primary Raynaud's disease (Wagner HH et al 1993) and stroke (Gainotti G, et al, 2001; Hayee Ma et al 2001), are associated with a high risk of depressive illness. So, NTG, being a disease involving vascular dysregulation, is postulated to be associated with psychopathology.

Glaucoma increases after 40 year-old and the number of people over this age in Hong Kong is rapidly growing. However, we have no knowledge about the link between psychopathology and NTG in Hong Kong. The present study is sought to overcome the limitation in previous research and the goals of present study are:

* To identify the prevalence of psychopathology of normal-tension glaucoma Hong Kong Chinese Out-patients attending a university-affiliated glaucoma clinic.
* To determine whether there are any differences among NTG patients, patients with glaucoma other than NTG and control in terms of psychopathology and quality of life.

Designs:

Case-control study to compare among patients with normal-tension glaucoma (NTG), patients with glaucoma other than normal-tension glaucoma (OTNTG) and control in terms of psychopathology and quality of life

DETAILED DESCRIPTION:
Patients with chronic medical illness have been shown to have higher rates of depression and other psychopathology (Kimmel PL et al, 1998; Amato L et al, 1996). Glaucoma is a chronic, progressive ophthalmologic disease. Treatment may involve the use of multiple medications and surgery. Despite therapy, many patients continue to worsen, and some may even lose vision. Because of this threat of potential loss of vision and the known depression-related side effects of some of topical glaucoma medication, particular beta-blocker (Cove-Smith JR et al, 1985), it can be necessary hypothesized that glaucoma patient may have an increased prevalence of depression and other psychopathology. It is also reasonable to apply similar hypothesis on the patients with normal-tension glaucoma.

Normal-tension glaucoma (NTG) is a type of open-angle glaucoma defined as an optic neuropathy with visual-field defects together normal distribution of intraocular pressure (<21 mmHg) over a period of twenty-four hour as well as normal chamber-angle anatomy (Levene RZ, 1980). NTG is associated with different vasospastic syndrome including higher incidence of migraine (Phelps CD et al, 1985), angina pectoris (Goldberg I et al, 1981), silent myocardial ischemia (Kaiser HJ et al, 1993) and ocular vasopasm (Flammer J et al, 1991; Flammer J et al 1987; Orgul S et al 1995). Such associated clinical characteristics suggest that the pathogenesis of NTG involves vascular dysregulation. In the past studies, it is well documented that many physical problems related to vascular dysregulation, such as angina pectoris (Friedman M et al 1974; Russek HI et al 1976), migraine (Diener HC et al 1994), primary Raynaud's disease (Wagner HH et al 1993) and stroke (Gainotti G, et al, 2001; Hayee Ma et al 2001), are associated with a high risk of depressive illness. So, NTG, being a disease involving vascular dysregulation, is postulated to be associated with psychopathology.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of patients (NTG and OTNTG):

* Cantonese-speaking Chinese
* Aged from 18 to 65
* Attending university-affiliated glaucoma clinic from August, 2005 to June, 2006 with written consent Inclusion criteria of control
* Those just receiving routine fundi examination without any ophthalmologic follow-up afterwards
* Cantonese-speaking Chinese
* Aged from 18 to 65
* With written consent

Exclusion Criteria of cases:

Exclusion criteria:

* Psychoses
* Psychiatric condition warranting hospitalization Exclusion criteria of control
* Previous or current ocular or general acute or chronic disease
* Taking any medication
* Psychoses
* Psychiatric condition warranting hospitalization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients from a tertiary University Ophthalmic clinic setting
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2006-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Karina Chan, MBChB, MRCPsych, Principal Investigator — Department of Psychiatry, Kowloon Hospital, Hong Kong; Dexter Leung, MBChB, FRCS, Study Director — Chinese University of Hong Kong; Sing Lee, MD, MRCPsych, Study Director — Department of Psychiatry, CUHK; Dennis Lam, MD, FRCOphth, Study Chair — Chinese University of Hong Kong
Locations (1):
- Department of Psychiatry, Kowloon Hospital, Hong Kong, Hong Kong, China